CLINICAL TRIAL: NCT04850573
Title: Effects of Equine Assisted Activities on Veterans With Post-traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Karyn Malinowski, Ph.D., Professor and Director, Rutgers Equine Science Center, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2019001999
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: veterans, equine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an equine assisted activities intervention or wait-listed control for eight weeks. At the end of the eight week period, participants assigned to the wait-listed control will be offered the opportunity to participate in the equine assisted activities intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAA (Experimental): Participants in this arm will take part in eight weekly thirty minute sessions of equine facilitated learning where they interact with a horse and learn basic horsemanship skills.
  Interventions: Other: equine assisted activities
- Control (No Intervention)

INTERVENTIONS:
Other: equine assisted activities — Participants interact with the horse and learn how to safely handle the horse.
  Other Names: equine facilitated learning, horsemanship
  Arms: EAA

SUMMARY:
The study will examine the effects of eight weeks of equine assisted activities (EAA) on co-regulation, basal physiological values, and symptom severity in veterans with post-traumatic stress disorder (PTSD). Heart rate, respiration rate, surface electromyography (EMG) and plasma concentrations of cortisol, epinephrine, norepinephrine, and oxytocin will be measured at rest and during dyadic interaction tasks (human to human or human to horse) to assess effects of EAA on these measures. Additionally, standard and regularly used questionnaires will be used to monitor PTSD symptom severity during the study and 6-month follow-up period. EAA is expected to lower PTSD symptom severity, and mitigate other physiological changes associated with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* male
* was deployed and experienced combat in Iraq or Afghanistan
* between 18 and 65 years of age

Exclusion Criteria:

* female
* amputation
* severe traumatic brain injury
* schizophrenia, bi-polar disorder, or substance dependence in the last 3 months
* pacemaker
* allergies to horses
* previous enrollment in equine assisted activities or psychotherapy in an equine environment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males are eligible for inclusion in the study because the hormones being measured are impacted by the menstrual cycle in females.
Enrollment: 9 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to the Conclusion of 8 weeks of EAA in PTSD Symptoms as Assessed by PCL-5 & Brief Symptom Inventory | Symptoms will be assessed prior to the intervention and immediately following the eight week intervention.
  The Brief Symptom Inventory and PTSD Checklist for DSM-5 are questionnaires used to assess the presence and severity of post-traumatic stress disorder symptoms.
Change from Baseline to 2-months After the Conclusion of EAA in PTSD Symptoms as Assessed by PCL-5 & Brief Symptom Inventory | Symptoms will be assessed prior to the intervention and 2-months after the end of the EAA sessions.
  The Brief Symptom Inventory and PTSD Checklist for DSM-5 are questionnaires used to assess the presence and severity of post-traumatic stress disorder symptoms.
Change from Baseline to 6-months After the Conclusion of EAA in PTSD Symptoms as Assessed by PCL-5 & Brief Symptom Inventory | Symptoms will be assessed prior to the intervention and 6-months after the end of the EAA sessions.
  The Brief Symptom Inventory and PTSD Checklist for DSM-5 are questionnaires used to assess the presence and severity of post-traumatic stress disorder symptoms.
Co-regulation of heart rate between horse and human during EAA sessions. | Co-regulation of heart rate between horse and human will be assessed once a week during a 30 min session for 8 weeks..
  Co-regulation will be assessed through the telemetric measurement and modeling of heart rate.
Co-regulation of cortisol between horse and human during EAA sessions. | Co-regulation of cortisol between horse and human will be assessed once a week during a 30 min session in weeks 1,4, and 8 of an 8 week period.
  Co-regulation will be assessed through collection of serial blood samples and subsequent measurement and modeling of plasma cortisol.
Co-regulation of oxytocin between horse and human during EAA sessions. | Co-regulation of oxytocin between horse and human will be assessed once a week during a 30 min session in weeks 1,4, and 8 of an 8 week period.
  Co-regulation will be assessed through collection of serial blood samples and subsequent measurement and modeling of plasma oxytocin.
Co-regulation of epinephrine between horse and human during EAA sessions. | Co-regulation of epinephrine between horse and human will be assessed once a week during a 30 min session in weeks 1,4, and 8 of an 8 week period.
  Co-regulation will be assessed through collection of serial blood samples and subsequent measurement and modeling of plasma epinephrine.
Co-regulation of norepinephrine between horse and human during EAA sessions. | Co-regulation of norepinephrine between horse and human will be assessed once a week during a 30 min session in weeks 1,4, and 8 of an 8 week period.
  Co-regulation will be assessed through collection of serial blood samples and subsequent measurement and modeling of plasma norepinephrine.
Co-regulation of muscle activity between horse and human during EAA sessions. | Co-regulation of muscle activity between horse and human will be assessed once a week during a 30 min session over an 8 week period.
  Co-regulation will be assessed through collection of surface electromyography (sEMG) from the masseter, brachiocephalas, and cervical trapezius muscles and subsequent modeling.
Changes in co-regulation of heart rate during dyadic (human-human) interactions following 8 weeks of EAA | Co-regulation will be assessed prior to the intervention and immediately following the eight week intervention.
  Co-regulation will be assessed through the measurement and modeling of heart rate during gazing, not looking, resting, and mimicking tasks.
Changes in social motor synchrony during dyadic (human-human) interactions following 8 weeks of EAA | Social motor synchrony will be assessed prior to the intervention and immediately following the eight week intervention.
  Social motor synchrony will be assessed through the measurement and modeling of gross motor movement during a pendulum swinging task.
Changes in resting heart rate following 8 weeks of EAA | Resting heart rate will be assessed prior to the intervention and immediately following the eight week intervention.
  Telemetric heart rate monitors will be used to collect resting heart rate.
Changes in basal plasma cortisol concentration following 8 weeks of EAA | Cortisol concentrations will be assessed prior to the intervention and immediately following the eight week intervention.
  Plasma concentrations of cortisol will be measured via immunoassay following blood draws during rest.
Changes in plasma basal oxytocin concentration following 8 weeks of EAA | Plasma oxytocin concentrations will be assessed prior to the intervention and immediately following the eight week intervention.
  Plasma concentrations of oxytocin will be measured via immunoassay following blood draws during rest.
Changes in basal plasma epinephrine concentration following 8 weeks of EAA | Plasma epinephrine concentrations will be assessed prior to the intervention and immediately following the eight week intervention.
  Plasma concentrations of epinephrine will be measured via immunoassay following blood draws during rest.
Changes in basal plasma norepinephrine concentration following 8 weeks of EAA | Plasma norepinephrine concentrations will be assessed prior to the intervention and immediately following the eight week intervention.
  Plasma concentrations of norepinephrine will be measured via immunoassay following blood draws during rest.

CONTACTS AND LOCATIONS:
Overall Officials: Karyn Malinowski, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Equine Science Center, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rankins EM, Quinn A, McKeever KH, Malinowski K. Ground-based adaptive horsemanship lessons for veterans with post-traumatic stress disorder: a randomized controlled pilot study. Front Psychiatry. 2024 May 28;15:1390212. doi: 10.3389/fpsyt.2024.1390212. eCollection 2024. PMID 38863605